CLINICAL TRIAL: NCT01861132
Title: Validation of Non-invasive Monitoring of Blood Pressure and Cardiac Output in Healthy Pregnant Women During Cesarean Section
Brief Title: Validation of a Non-invasive Hemodynamic Monitor (NexFin) in Pregnant Women
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Leiv Arne Rosseland, Head for R&D department, Oslo University Hospital
Other Study IDs: NexValid13
Record Dates: First submitted 2013-05-21; First posted 2013-05-23 (Estimated); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Hemodynamic Changes in Pregnancy
Keywords: Pregnancy, cesarean delivery, blood pressure, cardiac output

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy pregnant women: Healthy pregnant women for C-section under spinal anesthesia

SUMMARY:
Blood pressure and cardiac output can be measured invasively in pregnant women. Non-invasive monitoring devices are desirable, but until now, no equipment has proven validity. This study aims at validating the non-invasive monitoring device NexFin (second generation Finometer) in pregnant women.

DETAILED DESCRIPTION:
Validation will be a direct beat-to-beat comparison of data from NexFin and the invasive measurements of blood pressure and calibrated cardiac output as an integrated part of LiDCO Plus. Both comparison of absolute values and the two different devices trending abilities will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy singleton pregnancies at term scheduled for cesarean delivery

Exclusion Criteria:

* Twins, or multiple gestation, pre-eclampsia, gestational hypertension
* Reynaud phenomenon

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Healthy singleton pregnancies at term scheduled for cesarean delivery under spinal anesthesia
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2013-05; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Systolic blood pressure | 15 minutes
  Comparison of beat-to-beat data

SECONDARY OUTCOMES:
Cardiac output | 15 minutes
  Comparing beat-to-beat data of cardiac output

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital, Oslo, Norway

REFERENCES:
- [Result] Omenas IN, Tronstad C, Rosseland LA. Accuracy and trending abilities of finger plethysmographic blood pressure and cardiac output compared to invasive measurements during caesarean delivery in healthy women: an observational study. BMC Anesthesiol. 2020 Jun 27;20(1):157. doi: 10.1186/s12871-020-01078-8. PMID 32593297